CLINICAL TRIAL: NCT06338956
Title: Optimal Attained LDL-Cholesterol Levels in Patients Who Achieved ≥50% LDL Reduction After PCI
Acronym: Lipid-PCI
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Ki Hong Choi, Professor, Samsung Medical Center
Other Study IDs: Lipid-PCI
Record Dates: First submitted 2024-03-24; First posted 2024-04-01 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Coronary Artery Disease; Hyperlipidemias
Keywords: Percutaneous coronary intervention; Statin
MeSH Terms: conditions — Coronary Artery Disease; Hyperlipidemias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- >=50% LDL-C reduction: LDL-C reduction >=50%
  Further divided by LDL <55mg/dL 55< LDL < 70 mg/dL LDL > 70 mg/dL
  Interventions: Drug: LDL reduction therapy
- <50% LDL-C reduction: LDL-C reduction <50%
  Interventions: Drug: LDL reduction therapy

INTERVENTIONS:
Drug: LDL reduction therapy — LDL reduction therapy

SUMMARY:
For the management of low-density lipoprotein-cholesterol (LDL-C), some guidelines recommend initial statin treatment with high-intensity statins to achieve at least a 50% reduction in LDL-C levels. High-intensity or maximally tolerated intensity can be maintained without a target goal. However, the European guideline recommends less than 55 mg/dL of LDL-C after PCI.

DETAILED DESCRIPTION:
To investigate the Optimal Attained LDL-C Levels in Patients Who Achieved ≥50% LDL-C Reduction After PCI.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving PCI with health check up before and after PCI within 3 years

Exclusion Criteria:

* Patients receiving statin before PCI
* Patients with liver cirrhosis
* Patients with cancer
* Patients without prescription of statin
* Patients with LDL-C <55 mg/dL before PCI

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with coronary artery disease undergoing PCI
Sampling Method: Non-Probability Sample
Enrollment: 135877 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-05-15 (Actual)

PRIMARY OUTCOMES:
MACCE | 10 years after PCI
  major adverse cardiac and cerebrovascular events

SECONDARY OUTCOMES:
Cardiovascular death | 10 years after PCI
  death from cardiovascular cause
Spontaneous myocardial infarction | 10 years after PCI
  MI with hospitalziation
Repeat revascularization | 10 years after PCI
  additional PCI or CABG
Ischemic stroke | 10 years after PCI
  Stoke from ischemic cause

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kang D, Choi KH, Yang S, Kim H, Park TK, Lee JM, Cho J, Yang JH, Song YB, Choi SH, Gwon HC, Hahn JY. Clinical significance of low-density lipoprotein cholesterol percentage reduction and attained levels after percutaneous coronary intervention. CMAJ. 2025 Apr 27;197(16):E442-E452. doi: 10.1503/cmaj.241713. PMID 40294950